CLINICAL TRIAL: NCT01294098
Title: Examining the Efficacy of Femoral Nerve Block in Children With a Femoral Shaft Fracture
Brief Title: Efficacy Study of Femoral Nerve Block in Children With a Femur Fracture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients were not willing to be randomized and therefore recruitment could not continue.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-0331
Record Dates: First submitted 2011-02-09; First posted 2011-02-11 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Femoral Fractures; Pain, Postoperative
Keywords: Femoral Fractures; Pediatrics; Pain, Postoperative
MeSH Terms: conditions — Femoral Fractures; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PCA only (No Intervention): this group will only get a pain control anesthesia pump to use for post-operative pain
- PCA and femoral nerve block (Experimental): this group will be receiving a femoral nerve block during surgery and have a PCA post-operatively
  Interventions: Drug: Marcaine
- PCA + hematoma block (Experimental): patient will receive hematoma block during surgery
  Interventions: Drug: Marcaine

INTERVENTIONS:
Drug: Marcaine — 0.75 cc/kg of 1/4% Marcaine
  Other Names: bupivacaine
  Arms: PCA + hematoma block; PCA and femoral nerve block

SUMMARY:
The purpose of this study is to examine the efficacy of the use of Marcaine in femoral nerve blocks and hematoma blocks for post operative pain relief for femoral shaft fractures in a pediatric population.

DETAILED DESCRIPTION:
Children with femur fractures can have severe pain after elastic nail fixation. The current national standard for post operative pain control would be intravenous narcotics. In addition to the use of intravenous narcotics, there are two alternative methods used during the surgery in order to potentially decrease the pain post-operatively. These methods are hematoma block or a femoral nerve block. Both are proven safe and effective in children, however little research has been done to look at the effectiveness of these various methods compared to one another.

ELIGIBILITY:
Inclusion Criteria:

* A child with a femoral shaft fracture requiring surgical treatment and the placement of intramedullary nails
* Weight of 30-100 Kg
* Child must be older than 6 years old

Exclusion Criteria:

* Any child that had an open fracture
* A child that has a pain abnormality
* Any child with an allergy to local anesthetic
* Any child with a neurological injury
* Any child with the inability to report pain
* Any child that is unable to use a PCA post-operatively

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-10-08 (Actual); Study Completion 2014-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Eric Gordon, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - St. Louis Childrens Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PCA Only | PCA and Femoral Nerve Block | PCA + Hematoma Block
Started | 0 | 1 | 1
Completed | 0 | 0 | 0
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCA Only | PCA and Femoral Nerve Block | PCA + Hematoma Block | Total
Number analyzed (Participants) | 0 | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 1 | 1 | 2
  Between 18 and 65 years |  | 0 | 0 | 0
  >=65 years |  | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  | 13 [13 to 13] | 8 [8 to 8] | 10.5 [8 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0 | 0
  Male |  | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Scores
Description: We will be looking at post-operative pain scores to see if those in the intervention group have lower pains scores.
  Wong Baker FACES pain scale:The faces correspond to numeric values from 0-5. This scale can be documented with the numeric value. The pain scale goes from 0-5 with 0 being no pain and 5 being the worst pain.
  0: No Hurt
  1. Hurts a little bit
  2. Hurts a little more
  3. Hurts even more
  4. Hurts a whole lot
  5. Hurts worst
Time Frame: with in the first 24 hours
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | PCA Only | PCA and Femoral Nerve Block | PCA + Hematoma Block
Number analyzed (Participants) | 0 | 1 | 1
units on a scale |  | 1.1 [0 to 5] | .11 [0 to 1]

2. Primary Outcome: Post-operative Narcotic Use
Description: We will be looking at the amount of narcotics used after surgery to see if there is a reduction in narcotic use
Time Frame: within first 24 horus
Measure: Number; unit: mg
Arm/Group | PCA Only | PCA and Femoral Nerve Block | PCA + Hematoma Block
Number analyzed (Participants) | 0 | 1 | 1
mg |  | 14.4 | 3.2

3. Secondary Outcome: Femur Fracture Healing
Description: we will following patients to look at fracture healing post-operatively
Time Frame: first year
Measure: Number; unit: weeks
Arm/Group | PCA Only | PCA and Femoral Nerve Block | PCA + Hematoma Block
Number analyzed (Participants) | 0 | 1 | 1
weeks |  | 24 | 10

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | PCA Only | PCA and Femoral Nerve Block | PCA + Hematoma Block
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No